CLINICAL TRIAL: NCT03500302
Title: Effect of Evolocumab on Coronary Endothelial Function
Acronym: EVOLVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00127952
Record Dates: First submitted 2017-11-27; First posted 2018-04-18 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Human Immunodeficiency Virus; Coronary Artery Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Pilot clinical trial to study HIV+ patients with baseline coronary endothelial dysfunction and assess changes in that function from the baseline measure to 1 and 6 weeks following initiation of therapy with evolocumab so as to test the hypotheses that PCSK9 inhibition with evolocumab improves coronary endothelial function (CEF) measured directly and non-invasively with MRI at 1 week and 6 weeks after initiation of evolocumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Evolocumab (Experimental): All enrolled patients will receive evolocumab sq once a month for a total of two doses
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Evolocumab sq once a month for a total of two doses
  Other Names: Repatha

SUMMARY:
The investigators propose a pilot study using (1) MRI to assess coronary artery endothelial function, (2) brachial ultrasound to assess systemic endothelial function, (3) serum markers of inflammation and of endothelial cell function and (4) echocardiographic measures of left ventricular diastolic and systolic properties, before and following initiation of PCSK9 antibody in HIV positive subjects.

DETAILED DESCRIPTION:
To evaluate the effect of the PCSK9 inhibitor evolocumab on coronary and systemic endothelial function, systemic biomarkers of endothelial function and of inflammation, and echocardiographic measures of left ventricular diastolic and systolic properties in subjects who are HIV+. Potential participants will be asked to undergo a screening MRI exam. Those who have evidence of coronary endothelial dysfunction on the MRI exam will receive evolocumab 420 mg sq (the dose that is approved for treatment of hypercholesterolemia) following the screening exam and again at one month. Repeat MRI and ultrasound measures of coronary and systemic endothelial function, as well as serum markers of endothelial function and inflammation, and echocardiographic measures of diastolic and systolic left ventricular function will be obtained at one and six weeks following the first administration of evolocumab.

The investigators will test the hypotheses that PCSK9 inhibition improves endothelial function measured non-invasively on MRI and systemic markers of inflammation at one week (+/- 3 days) and six weeks after initiation of the PCSK9 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Participants of either gender who are >21 years of age (no upper age limit)
* HIV (Human Immunodeficiency Virus) positive and taking stable Anti-Retroviral Therapy (ART), no change in regimen in last 3 months)
* Undetectable HIV viral load (plasma HIV RNA concentration, RNA=Ribonucleic Adic)
* Abnormal coronary endothelial function on MRI (Magnetic Resonance Imaging) at baseline (<5% change in coronary cross sectional area during isometric handgrip exercise as compared to resting value).
* Lipids at screening visit: Fasting LDL-C >70 mg/dL (LDL-C=Low Density Lipoprotein Cholesterol); fasting TG<500 mg/dL (TG=Triglycerides)
* Permission of treating physician

Exclusion Criteria:

* Patients unable to understand the risks, benefits, and alternatives of participation and give meaningful consent.
* Patients with contraindications to MRI such as implanted metallic objects (pre-existing cardiac pacemakers, cerebral clips),
* History of a recent cardiovascular or cerebrovascular events or procedure (e.g. myocardial infarction, stroke, transient ischemic attack, angioplasty, Coronary artery bypass surgery) during the past 90 days.
* Subjects with prior exposure to evolocumab or another PCSK9 (Proprotein convertase subtilisin/kexin type 9) inhibitor.
* Pregnant women or breastfeeding women. Women of childbearing potential (even if using oral contraceptive agents) or intention to breastfeed.
* History of alcoholism or drug addiction according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria within 12 months prior to screening. Use of any recreational drugs within 6 months prior to screening.
* Renal impairment defined by estimated glomerular filtration rate <45 ml/min.
* Moderate-severe hepatic disease (elevation in hepatic transaminases >3x upper limit of normal, ULN) or direct bilirubin >3.0 X ULN at screening.
* Cluster of differentiation 4 (CD4)<200 cell/mm3
* Congestive heart failure, New York Heart Association functional class III or greater, or left ventricular ejection fraction measured by imaging known to be <30%. (Imaging not required for study inclusion).
* History of allergic or anaphylactic reaction to any therapeutic monoclonal antibody (IgG protein) or molecules made of components of monoclonal antibodies
* Active phase hepatitis. Stable patients with hepatitis B or C infection >3 years before randomization are eligible.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Hays, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leucker TM, Gerstenblith G, Schar M, Brown TT, Jones SR, Afework Y, Weiss RG, Hays AG. Evolocumab, a PCSK9-Monoclonal Antibody, Rapidly Reverses Coronary Artery Endothelial Dysfunction in People Living With HIV and People With Dyslipidemia. J Am Heart Assoc. 2020 Jul 21;9(14):e016263. doi: 10.1161/JAHA.120.016263. Epub 2020 Jul 17. PMID 32674634

RESULTS

PARTICIPANT FLOW:
Groups:
- Evolocumab: All enrolled patients (people living with HIV) who received evolocumab sq once a month for a total of two doses
Period: Overall Study
Arm/Group | Evolocumab
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Evolocumab Group: Patients (people living with HIV) who received Evolocumab sq once a month for total of 2 doses
Arm/Group | Evolocumab Group
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26 (5)

OUTCOME MEASURES:

1. Primary Outcome: Coronary Endothelial Function as Assessed by Percent Coronary Artery Area Change With Isometric Handgrip Exercise
Description: Coronary endothelial function will be assessed by the percent change in cross sectional coronary artery area (measured on MRI) from rest to isometric handgrip stress exercise at week 1 and week 6. The percent change from week 1 to week 6 is presented below.
Time Frame: 1 week and 6 weeks
Measure: Mean (Standard Deviation); unit: percent change in coronary artery area
Groups:
- Evolocumab: Patients with HIV receiving Evolocumab sq (2 doses total)
Arm/Group | Evolocumab
Number analyzed (Participants) | 19
percent change in coronary artery area | 5.6 (5.5)

2. Secondary Outcome: LDL Cholesterol Level
Description: LDL cholesterol level: mg/dL.
Time Frame: At 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Evolocumab
Number analyzed (Participants) | 19
mg/dL | 37 (19)

ADVERSE EVENTS:
Time Frame: Up to 10 weeks from start of study.
Groups:
- Evolocumab: All enrolled patients who received evolocumab sq once a month for a total of two doses.
Arm/Group | Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03500302/Prot_SAP_000.pdf